CLINICAL TRIAL: NCT02508792
Title: Acute Effects of Low Level Laser Therapy in Muscle Function of Patients With Heart Failure.
Brief Title: Low Level Laser Therapy in Heart Failure Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Pedro Dal Lago, Doctor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 37904814.0.0000.5345
Record Dates: First submitted 2015-07-22; First posted 2015-07-27 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LASER (Active Comparator): Subject will receive application of LASER before muscle fatigue protocol.
  Note: this is a crossover study.
  Interventions: Device: LASER
- LASER PLACEBO (Placebo Comparator): Subject will receive application of LASER (now deactivated) before muscle fatigue protocol.
  Note: this is a crossover study.
  Interventions: Device: LASER PLACEBO

INTERVENTIONS:
Device: LASER — Low level LASER therapy will be applied in six different regions of the thight from the dominant limb, before a fatigue protocol using a isokinetic equipment.
  Arms: LASER
Device: LASER PLACEBO — The low level LASER therapy turned off (placebo) will be applied in six different regions of the thight from the dominant limb, before a fatigue protocol using a isokinetic equipment.
  Arms: LASER PLACEBO

SUMMARY:
Heart failure (HF) is an important public health problem being considered an emerging epidemic, therefore, strategies are essential to improve symptoms and to decrease the money expenditure on healthcare. Based on the knowledge about the syndrome of heart failure, new approaches are needed to decrease the symptoms, to enhance the quality of life of these patients and highlight the non-pharmacological therapies such as the use of phototherapy. The objective of this study is to study the effect of low level laser therapy in muscle function and tissue oxygenation of the lower limbs in patients with heart failure. It is a randomized, double-blind, including 20 individuals with heart failure, with stable, class II or III according to the New York Heart Association (NYHA). It will be evaluated the acute effects of a LASER intervention applied before a fatigue protocol throught muscle function and tissue oxygenation in the participants. Evaluations will be performed by an isokinetic dynamometer, near infrared spectroscopy (NIRS) and electromyography . It will be analyzed the concentration of oxyhemoglobin and deoxyhemoglobin, total hemoglobin concentration, the difference between these concentrations, muscular torque, fatigue index and muscle activation. The data will be subjected to distribution normality test and if they have normal distribution, the differences between the interventions will be checked by analysis of variance, considering significant ap <0.05. If the data is non-parametric distribution will be using the Mann-Whitney or Kruskal-Wallis. The SPSS 19.0 software will be used as a tool for data analysis. The investigators expected to find as outcomes of this study an increase in peripheral muscle function and tissue oxygenation and also a delay in the development of muscle fatigue in patients with HF submitted to acute intervention with LASER.

DETAILED DESCRIPTION:
Day 1: Informed Consent signature and Clear (IC); Application of the Minnesota Living with Heart Failure Questionnaire (MLHFQ); Measurement of the muscle thickness with use of ultrasound; Anatomical points definition for electrode placement of Electromyography (EMG); Warming up on stationary bike; Subject's position in the Isokinetic, placement of EMG electrodes and NIRS´ optodes; Baseline measurement (peak torque and muscle fatigue protocol); Stretching exercises for the lower limbs muscles; 48-hour interval.

Day 2: Warming up on stationary bike; LASER / Placebo application; Subject's position in the Isokinetic, placement of EMG electrodes and NIRS´ optodes; Peak torque and muscle fatigue protocol in the Isokinetic equipment; Stretching exercises for the lower limbs muscles; 48-hour interval.

Day 3: Warming up on stationary bike; LASER / Placebo application; Subject's position in the Isokinetic, placement of EMG electrodes and NIRS´ optodes; Peak torque and muscle fatigue protocol in the Isokinetic equipment; Stretching exercises for the lower limbs muscles.

ELIGIBILITY:
Inclusion Criteria:

* Participants who consent to cooperate with this study and meet the following inclusion criteria: a) to have a clinical diagnosis of heart failure (ejection fraction of the left ventricle less than 40% secondary to ischemia or idiopathic dilated cardiomyopathy) functional class II or III, according to the NYHA classification ; b) be medically stable in the 30 days prior to enrollment in the study and, c) not have participated or are participating in cardiac rehabilitation program.

Exclusion Criteria:

* The sample shall be excluded: a) participants who did not consent to participate in the study, b) participants with present insufficient level of understanding for the tests, c) participants that are making use of anti-inflammatory drugs steroids and nonsteroidal, d) the ones that have limitations to perform physical activity (exacerbation of fatigue, extreme breathlessness, arthritis, claudication, angina), e) participants with musculoskeletal disease, brain vascular disease and psychiatric illness and f) the ones who not adhere to the schedule of activities proposed in the study.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in muscle torque after a fatigue protocol in HF patients | 8 days
  Muscle torque with an isokinetic equipment will be accessed after a fatigue protocol in patients with heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Dal Lago, Doctor, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- UFCSPA, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Albuquerque-Pontes GM, Vieira RP, Tomazoni SS, Caires CO, Nemeth V, Vanin AA, Santos LA, Pinto HD, Marcos RL, Bjordal JM, de Carvalho Pde T, Leal-Junior EC. Effect of pre-irradiation with different doses, wavelengths, and application intervals of low-level laser therapy on cytochrome c oxidase activity in intact skeletal muscle of rats. Lasers Med Sci. 2015 Jan;30(1):59-66. doi: 10.1007/s10103-014-1616-2. Epub 2014 Jun 24. PMID 24957189
- [Background] Baroni BM, Leal Junior EC, De Marchi T, Lopes AL, Salvador M, Vaz MA. Low level laser therapy before eccentric exercise reduces muscle damage markers in humans. Eur J Appl Physiol. 2010 Nov;110(4):789-96. doi: 10.1007/s00421-010-1562-z. Epub 2010 Jul 3. PMID 20602109
- [Background] Blum A. Heart failure--new insights. Isr Med Assoc J. 2009 Feb;11(2):105-11. PMID 19432040
- [Background] Carvalho VO, Guimaraes GV, Carrara D, Bacal F, Bocchi EA. Validation of the Portuguese version of the Minnesota Living with Heart Failure Questionnaire. Arq Bras Cardiol. 2009 Jul;93(1):39-44. doi: 10.1590/s0066-782x2009000700008. English, Portuguese, Spanish. PMID 19838469
- [Background] Conraads VM, Van Craenenbroeck EM, De Maeyer C, Van Berendoncks AM, Beckers PJ, Vrints CJ. Unraveling new mechanisms of exercise intolerance in chronic heart failure: role of exercise training. Heart Fail Rev. 2013 Jan;18(1):65-77. doi: 10.1007/s10741-012-9324-0. PMID 22684340
- [Background] Leal Junior EC, Lopes-Martins RA, Dalan F, Ferrari M, Sbabo FM, Generosi RA, Baroni BM, Penna SC, Iversen VV, Bjordal JM. Effect of 655-nm low-level laser therapy on exercise-induced skeletal muscle fatigue in humans. Photomed Laser Surg. 2008 Oct;26(5):419-24. doi: 10.1089/pho.2007.2160. PMID 18817474
- [Background] Lima A, Bakker J. Near-infrared spectroscopy for monitoring peripheral tissue perfusion in critically ill patients. Rev Bras Ter Intensiva. 2011 Sep;23(3):341-51. English, Portuguese. PMID 23949407
- [Background] Neves EB, et al. Comparação do percentual de gordura obtido por bioimpedância, ultrasson e dobras cutâneas em adultos jovens. Rev Bras Med Esporte 19(5): 323-327, 2013.
- [Background] Rondelli RR, Dal Corso S, Simoes A, Malaguti C. Methods for the assessment of peripheral muscle fatigue and its energy and metabolic determinants in COPD. J Bras Pneumol. 2009 Nov;35(11):1125-35. doi: 10.1590/s1806-37132009001100011. English, Portuguese. PMID 20011849